CLINICAL TRIAL: NCT02372591
Title: Analgesic Effects and Abuse Liability of Intravenous Hydromorphone and Buprenorphine in Opioid Dependent Participants With Chronic Musculoskeletal Pain
Brief Title: Study of the Treatment of Experimental Pain in Buprenorphine Maintained Persons With Chronic Musculoskeletal Pain
Acronym: 1401
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00093537; K23DA029609 (NIH)
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Opioid-Related Disorders; Chronic Pain
Keywords: Quantitative Sensory Testing; Hydromorphone; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination; Hydromorphone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Hydromorphone (Active Comparator)
  Interventions: Drug: Hydromorphone
- Buprenorphine (Experimental)
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Intravenous injection of approximately 10 mL administered via slow push over 5 minutes. Given 4 injections during the session with each injection separated by 1.5 hours.
  Other Names: Suboxone; Subutex
  Arms: Buprenorphine
Drug: Hydromorphone — Intravenous injection of approximately 10 mL administered via slow push over 5 minutes. Given 4 injections during the session with each injection separated by 1.5 hours.
  Other Names: Dilaudid
  Arms: Hydromorphone
Drug: Placebo — Intravenous injection of approximately 10 mL administered via slow push over 5 minutes. Given 4 injections during the session with each injection separated by 1.5 hours.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Pain is very common in persons with a history of addiction, but few studies have examined the best treatment of pain in this population. This is a study to determine the pain relief provided by intravenous hydromorphone (Dilaudid) or buprenorphine given to persons maintained on stable doses of methadone or buprenorphine who have chronic musculoskeletal pain. Experimental sessions will require overnight stays on a residential research unit. In these sessions, persons will be exposed to standard experimental pain techniques at baseline and then rate the relief (if any) provided by the study medication when exposed to the same techniques. Persons will be asked to participate in 3 sessions, each separated by at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

Opioid dependence according to the Mini International Neuropsychiatric Interview (MINI) and verified by the PI; urine toxicology negative for drugs of abuse but positive for opioid maintenance agent; stable buprenorphine (12-16 mg) dose for the past 30 days; chronic musculoskeletal pain (>3 months) as documented in medical history and physical; able and willing to perform/tolerate pain procedures; able to communicate in English.

Exclusion Criteria:

Current illicit substance use at screening or during trial as verified by urine toxicology screen and/or self-report (including cannabis use); current alcohol dependence as assessed on the MINI); medical or psychiatric condition known to influence quantitative sensory testing (QST) (e.g. HIV, peripheral neuropathy, current Major Depressive Disorder, Schizophrenia, Raynaud's syndrome); use of prescribed or over the counter analgesic agents or psychotropic medications known to have analgesic properties for 24 hours prior to session; previous allergic reaction to hydromorphone or buprenorphine; women who are pregnant, lactating or planning to get pregnant during the course of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Cold pressor test | This will be measured 7 times during each 40-hour session. On average, all sessions will be completed within 4 weeks.
  The participant places a hand up to the wrist in a circulating water bath maintained at approximately 4 degrees Celsius (up to 5 minutes). The time at which pain develops is the threshold. The time a volunteer's hand remains underwater before pain is unbearable is tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: D. Andrew Tompkins, M.D. M.H.S., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States